CLINICAL TRIAL: NCT04533711
Title: Physical Activity Pathway for Patients With Osteoarthritis in Primary Care
Brief Title: Physical Activity Pathway for Patients With Osteoarthritis in Primary Care (OA-PCP) (R33)
Acronym: OA-PCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-2134; 4R33AG056568-03 (NIH)
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA-PCP (Experimental): Participants assigned to the OA-PCP intervention will receive an initial physical activity (PA) coaching call then, 5 more calls over the course of 12 months. Participants, if they agree, will also receive monthly check-in emails between phone calls.
  Interventions: Behavioral: OA-PCP Intervention
- Attention Control (Placebo Comparator): Participants assigned to the Attention Control group will receive the same number of phone calls over the course of 12 months, focused on understanding osteoarthritis (OA) and current information on treatment options. Participants, if they agree, will also receive monthly check-in emails between phone calls.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: OA-PCP Intervention — The OA-PCP intervention includes brief physical activity (PA) counseling delivered via phone by a PA Coach trained in relevant aspects of PA and motivational interviewing. During the initial call, the PA Coach will ask participants about their current physical activity level and work with them to set physical activity goals. Then, after the first call, participants in this group will receive a call about two weeks later, then at about 3 months, 6 months, 9 months and 12 months later. During these calls, the PA coach will ask participants' about their progress toward PA goals and work with them to address any barriers or challenges. The coach will also help participants to identify any programs or resources that may help them to achieve their PA goals. Participants in this group will be asked to wear a wrist-worn monitor to help them track their PA during the intervention period. Also, if participants approve, the coach will use an online program to view their PA data.
  Arms: OA-PCP
Behavioral: Attention Control — This group will receive an intervention in the same "dose" (e.g., number and duration of phone calls and emails) as the OA-PCP group, but the content will not be PA-specific. During the first call, the Coach will discuss 2 topics, for which the amount of content parallels call #1 for the OA-PCP: What is OA? OA Diagnosis and OA Risk Factors. During the second call, the Coach will discuss the topic of Health Care Providers and Overview of OA Treatment Guidelines. Call topics for 3, 6, 9 and 12- month follow-up calls will be: Pain Medications, Mechanical Treatments (e.g., knee braces, footwear, joint protection), Complimentary and Alternative Therapies and discussion of OA and Mental Health, Sleep and Fatigue.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to test an osteoarthritis (OA) primary care Physical activity Care Pathway (OA-PCP), a scalable intervention that includes: 1) a practical process for physical inactivity screening in primary care, 2) a brief, tailored physical activity (PA) counseling intervention via telephone, 3) connection of patients with community programs and other resources to support PA, and 4) follow-up with patients to deliver additional appropriate counseling and referrals to PA resources. This program will be compared to another program that provides education on a variety of topics important to understanding osteoarthritis (OA) and its care.

DETAILED DESCRIPTION:
This study will be a randomized pilot trial of the refined OA-PCP among n=240 patients age ≥65 with hip and/or knee OA recruited from primary care clinics. Participants will be assigned equally to either the OA-PCP or an attention control group. Participants will complete assessments at baseline, and 6-month and 12-month follow-up. Primary endpoint of the trial will be objectively assessed PA, measured via accelerometer and secondary endpoint will be self-reported pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* One other chronic health condition that qualified under Chronic Care Management (CCM) guidelines, including: diabetes, depression, hypertension, hyperlipidemia, heart failure, atrial fibrillation, ischemic heart disease, stroke/transient ischemic attack (TIA), peripheral vascular disease, Chronic obstructive pulmonary disease (COPD), bronchiectasis, asthma, rheumatoid arthritis, osteoarthritis, HIV/AIDS, chronic kidney disease, hepatitis (chronic & viral B & C) and osteoporosis
* Current Joint Symptoms
* Self-reported physical activity <150 minutes per week
* Willing to make a change in PA over the next 3 months

Exclusion Criteria:

* Pain in chest when performing physical activity
* Pain in chest when not performing physical activity
* Loss of balance because of dizziness or loss of consciousness
* Recommendation from doctor to only perform physical activity under medical supervision
* No documented diagnosis of knee or hip OA
* Dementia or other memory loss condition
* Active diagnosis of psychosis
* Active Substance abuse disorder
* Total knee or hip replacement surgery, meniscus tear, ligament tear, or other significant lower extremity injury or surgery in the last 6 months
* Severe hearing or visual impairment
* Serious/terminal illness as indicated by referral to hospice or palliative care
* Unstable angina
* Hospitalization for cardiovascular event in last 6 months
* History of ventricular tachycardia
* Unstable chronic obstructive pulmonary disease (2 hospitalizations within the previous 6 months and/or on oxygen)
* Stroke with moderate to severe aphasia
* Recent history (last 6 months) of three or more falls

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/ sharing agreement with University of North Carolina at Chapel Hill (UNC).
Supporting Information: SAP
Time Frame: Data will become available following publication of primary and secondary outcomes. Research study records will be maintained for no less than 6 years following the completion of the study.
Access Criteria: Data will be accessible following publication of study results and will be available for no less than 6 years following the completion of the study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OA-PCP | Attention Control
Started | 120 | 120
Completed 6-month Assessments | 92 | 102
Completed 12-month Assessments | 87 | 95
Completed | 87 | 95
Not Completed | 33 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OA-PCP | Attention Control | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.88 (4.79) | 73.56 (4.86) | 73.22 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 98 | 199
  Male | 19 | 22 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 117 | 115 | 232
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 38 | 74
  White | 82 | 77 | 159
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 6 in Objectively Assessed Physical Activity (Accelerometer)
Description: Minutes of moderate to vigorous intensity physical activity (MVPA) per week measured via accelerometer
Time Frame: Baseline, Month 6 (Follow-up)
Population: 46 participants did not complete 6-month follow-up assessments, and 30 did not have adequate physical activity data for this measure.
Measure: Mean (95% Confidence Interval); unit: Minutes per week
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 84 | 80
Minutes per week | -2.40 [-13.6 to 8.78] | -10.8 [-22.1 to 0.58]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.3086, Mixed Models Analysis; Mean Difference (Final Values) = 8.35, 95% CI 2-sided [-7.68 to 24.38]

2. Primary Outcome: Change From Baseline to Month 12 for Minutes in Objectively Assessed Physical Activity (Accelerometer)
Description: Minutes of moderate to vigorous intensity physical activity (MVPA) per week measured via accelerometer
Time Frame: Baseline, Month 12 (Follow-up)
Population: 58 participants did not complete 12-month follow-up assessments, and 26 did not have adequate physical activity data for this measure.
Measure: Mean (95% Confidence Interval); unit: Minutes per week
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 72 | 84
Minutes per week | 1.72 [-9.91 to 13.36] | -9.21 [-20.0 to 1.61]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.1820, Mixed Models Analysis; Mean Difference (Final Values) = 10.93, 95% CI 2-sided [-5.06 to 26.92]

3. Secondary Outcome: Change From Baseline to Month 6 for Steps Per Day
Description: Step counts measured via an accelerometer device.
Time Frame: Baseline, Month 6 (Follow-up)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 84 | 80
steps per day | -1.00 [-252 to 249.6] | -309 [-563 to -56.2]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.094, Mixed Models Analysis; Mean Difference (Final Values) = 308.4, 95% CI 2-sided [-50.2 to 667.1]

4. Secondary Outcome: Change From Baseline to Month 12 for Steps Per Day
Description: Step counts measured via an accelerometer device.
Time Frame: Baseline, Month 12 (Follow-up)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 72 | 84
steps per day | -80.9 [-356 to 193.8] | -433 [-689 to -177]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.0691, Mixed Models Analysis; Mean Difference (Final Values) = 352.0, 95% CI 2-sided [-25.2 to 729.2]

5. Secondary Outcome: Change From Baseline to Month 6 for Minutes of Sedentary Activity
Description: Minutes of sedentary activity measured via an accelerometer device.
Time Frame: Baseline, Month 6 (Follow-up)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 84 | 80
minutes per day | 0.26 [-11.5 to 11.98] | 6.11 [-5.78 to 18.00]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.4953, Mixed Models Analysis; Mean Difference (Final Values) = -5.85, 95% CI 2-sided [-22.6 to 10.94]

6. Secondary Outcome: Change From Baseline to Month 12 for Minutes of Sedentary Activity
Description: Minutes of sedentary activity measured via an accelerometer device.
Time Frame: Baseline, Month 12 (Follow-up)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 72 | 84
minutes per day | 8.05 [-4.89 to 20.98] | 10.30 [-1.72 to 22.31]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.8041, Mixed Models Analysis; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-20.0 to 15.49]

7. Secondary Outcome: Change From Baseline to Month 6 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Function Subscale
Description: The Western Ontario and McMasters Universities Osteoarthritis (WOMAC) function subscale includes 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty), with ranges of 0-68 for the function subscale with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Month 6 (Follow-up)
Population: 46 participants did not complete 6-month follow-up assessments, and 2 did not have adequate data for this measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 92 | 100
score on a scale | -1.06 [-3.15 to 1.04] | -1.12 [-3.13 to 0.89]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.9645, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-2.86 to 2.99]

8. Secondary Outcome: Change From Baseline to Month 12 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Function Subscale
Description: as for outcome 7
Time Frame: Baseline, Month 12 (Follow-up)
Population: 58 participants did not complete 12-month follow-up assessments, and 4 did not have adequate data for this measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 85 | 93
score on a scale | -2.95 [-5.22 to -0.67] | -0.27 [-2.44 to 1.91]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.0989, Mixed Models Analysis; Mean Difference (Final Values) = -2.68, 95% CI 2-sided [-5.85 to 0.49]

9. Secondary Outcome: Change From Baseline to Month 6 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale
Description: The Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale is a measure of lower extremity pain. It includes 5 items rated on a Likert scale of 0 (no pain) to 4 (extreme pain), with a total range of 0-20 with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Month 6 (Follow-up)
Population: 46 participants did not complete 6-month follow-up assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 92 | 102
score on a scale | -0.56 [-1.22 to 0.09] | -0.70 [-1.33 to -0.08]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.7667, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.77 to 1.05]

10. Secondary Outcome: Change From Baseline to Month 12 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale
Description: as for outcome 9
Time Frame: Baseline, Month 12 (Follow-up)
Population: 58 participants did not complete 12-month follow-up assessments.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OA-PCP | Attention Control
Number analyzed (Participants) | 87 | 95
score on a scale | -1.39 [-2.11 to -0.68] | -0.52 [-1.21 to 0.16]
Statistical Analysis 1: Comparison: OA-PCP vs Attention Control; Test type: Superiority; p = 0.0894, Mixed Models Analysis; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.87 to 0.13]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | OA-PCP | Attention Control
All-Cause Mortality (participants affected / at risk) | 1/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 1/120 | 0/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OA-PCP (N=120) | Attention Control (N=120)
Neurological symptoms (Nervous system disorders) | 1 (1) | 0 (0) — Patient presented to the emergency department complaining of dizziness, a feeling of pressure of the left arm, visual disturbances, chills, fatigue, headaches, nausea, and bilateral tingling of the feet and right arm. Patient was not hospitalized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT04533711/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04533711/ICF_000.pdf